CLINICAL TRIAL: NCT03562754
Title: Randomized Controlled Trial of Intermittent Hemodialysis With Regional Citrate Anticoagulation Versus Systemic Low Dose Heparin Anticoagulation in Patients at Risk of Bleeding in Nephrology Intensive Care Unit
Brief Title: Control Trial of Intermittent Hemodialysis With Regional Citrate VS Priming Heparin With Predilution in Patients at Risk of Bleeding
Acronym: ROBIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/NIMAO2/OM-01; 2018-A00141-54 (Other: ANSM)
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2020-11

CONDITIONS: Hemodialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Procedure: reduced systemic heparin anticoagulation
- Prometheus System (Experimental)
  Interventions: Procedure: Regional Citrate Anticoagulation

INTERVENTIONS:
Procedure: reduced systemic heparin anticoagulation — receive intermittent hemodialysis (Frésenius 4008) with blood flow at least of (200 ml/min) with double vascular access, biocompatible membrane dialyzer, low dose non fractionated heparine (5000 UI initially) and predilution with 25 mls/min dialysate
  Arms: Control
Procedure: Regional Citrate Anticoagulation — intermittent hemodialysis using Prometheus System with blood flow at least of 200 ml/min with double vascular access, biocompatible membrane dialyzer
  Arms: Prometheus System

SUMMARY:
The study investigators hypothesize that intermittent hemodialysis with regional citrate anticoagulation (Prometheus system/Frésénius) is more efficient than reduced systemic heparin anticoagulation in patients at bleeding risk hospitalized in nephrology intensive care unit

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed.
* The patient must have given his/her informed and signed consent.
* The legal guardian or trusted-person of an adult under guardianship must have given their informed and signed consent.
* The patient has health insurance coverage via the French social security system.
* The patient is at least 18 years old.
* The patient is at bleeding risk; the bleeding risk is defined by the clinical situation and according to predefined clinical situations (before or after surgery or biopsy, hemorrhage).
* The patient requires an intermittent hemodialysis in a nephrology ICU setting.

Exclusion Criteria:

* The patient is participating in, or has participated in over the past three months, another interventional trial.
* The patient is in an exclusion period determined by a previous study.
* The patient is under judicial protection.
* The parents (or legal guardian) of the patient refuse to sign the consent.
* It is impossible to correctly inform the patient/parents (or legal guardian) of the patient (language barrier).
* Contraindication to heparin treatment.
* Indication of continuous dialysis in ICU.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Duration of intermittent hemodialysis between groups | End of intermittent hemodialysis session (average 4 hours)
  Minutes

SECONDARY OUTCOMES:
Hemodialysis treatment adequacy | End of intermittent hemodialysis session (average 4 hours)
  KT/V value
Transmembrane pressure between groups | End of intermittent hemodialysis session (average 4 hours)
Blood aspect in the extracorporeal treatment circuit | End of intermittent hemodialysis session (average 4 hours)
  Clotting phenomena
Occurrence of hemorrhage | Hour 12
  Yes/no
Occurrence of metabolic disorders (hypocalcemia, metabolic alkalose) | Hour 12
  Yes/no
Occurance of unexpected complications (almost none recorded in the literature) | End of intermittent hemodialysis session (average 4 hours)
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moranne, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Faguer S, Serre JE, Brusq C, Bongard V, Casemayou A, Moranne O, Pfirmann P, Rafat C, Cointault O. A randomized crossover trial of regional anticoagulation modalities for intermittent haemodialysis. Nephrol Dial Transplant. 2025 Feb 28;40(3):537-543. doi: 10.1093/ndt/gfae155. PMID 38977911